CLINICAL TRIAL: NCT05688358
Title: Serum Interleukin - 17A in Juvenile Idiopathic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat-Allah Khaled Tolba Abdelraheem, Resident doctor, Assiut University
Other Study IDs: Interleukin - 17A in JIA
Record Dates: First submitted 2023-01-07; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: JIA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum levels of interleukin-17A in JIA — IL17 A by Enzyme linked immunosorbent assay method

SUMMARY:
1. This study aims to determine the serum levels of interleukin-17A (IL-17A) in children with juvenile idiopathic arthritis (JIA)
2. Analyze the correlation between IL-17A values and disease activity, certain clinical features, and laboratory markers of inflammation.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) is a group of chronic heterogenous disorders that manifests as joint inflammation in patients aged <16 years and lasts longer than 6 weeks. Globally, approximately 3 million children and young adults are suffering from JIA with prevalence rates consistently higher in girls. The prevalence of JIA in Africa and Middle East was observed to be towards the lower range of the global estimate. (1) The precise cause and pathogenesis of JIA are unknown; however, genetic, environmental, and autoimmune factors are hypothesized to play a role in its development. (2) The condition can affect one or more joints and cause systemic symptoms such as fever or rash, as well as extra-articular inflammatory signs such as uveitis.(3)

The IL-17 cytokine superfamily is composed of 6 structurally related cytokines, namely IL-17A-F. The most investigated member of the family is IL-17A. It is synthesized by Th17 cells, γδ-T cells, NK T cells, lymphoid tissue inducer-like cells, Paneth cells, and neutrophils. IL-17A plays important roles in protection from bacterial and fungal infections and in the development of autoimmune diseases (4)

Recently, a number of studies have been conducted on the role of IL-17A in the development of chronic arthritis. It has a role both at the initial stages of joint inflammation and in the destruction of joint cartilage and bone structures.(5) It binds to its receptors on synoviocytes, endothelial cells, fibroblasts and osteoblasts and stimulates production of pro-inflammatory cytokines, chemokines and other inflammatory mediators, and also, interacts synergistically with other pro- inflammatory cytokines such as IL-1, IL-6, and tumor necrosis factor alpha.(6)

ELIGIBILITY:
Inclusion Criteria:_ Patients less than 16 years at onset of disease and diagnosed with oligoarticular and polyarticular JIA, fulfilling the ILAR classificationcriteria of JIA.

* Control group will include age-and-sex-matched apparently healthy children.

Exclusion Criteria: • Patients having associated neurological or disabling diseases.

* Patients with diabetes mellitus, acute or chronic infections.
* Patients with another causes of arthritis other than JIA.

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: Patients less than 16 years at onset of disease and diagnosed with oligoarticular and polyarticular JIA, fulfilling the ILAR classificationcriteria of JIA.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Serum Interleukin - 17A in juvenile idiopathic Arthritis | baseline
  This study aims to determine the serum levels of interleukin-17A (IL-17A) in children with juvenile idiopathic arthritis (JIA)
  -Analyze the correlation between IL-17A values and disease activity, certain clinical features, and laboratory markers of inflammation

REFERENCES:
- See also: Interleukin-17A Levels Increase in Serum of Children With Juvenile Idiopathic — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6190946/